CLINICAL TRIAL: NCT01256736
Title: Prospective, Open-labeled, 1 Year Extension Study of the Efficacy and the Safety During Treatment of Tocilizumab in Patients With Active RA Completing Treatment CWP-TCZ301 Study
Brief Title: To Evaluate 1 Year Extension Study of the Efficacy and Safety of Tocilizumab in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWP-TCZ302
Record Dates: First submitted 2010-10-28; First posted 2010-12-09 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Antirheumatic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tocilizumab 8mg/kg + DMARDs (Experimental)
  Interventions: Drug: Tocilizumab; Drug: DMARDs

INTERVENTIONS:
Drug: Tocilizumab — intravenously at dose of 8mg/kg over 1 hour infusion every 4weeks
Drug: DMARDs — DMARDs(chloroquine, hydroxychloroquine, parenteral gold, sulfasalazine, azathioprine, and leflunomide)

SUMMARY:
The purpose of this study is to evaluate 1 year extension study of the efficacy and the safety during treatment tocilizumab in patients completing treatment CWP-TCZ301 study with moderate to severe active RA and an inadequate response to current DMARD.

ELIGIBILITY:
Inclusion Criteria:

* Patients Who have been satisfied the in/exclusion criteria of CWP-TCZ301
* Patients who have been withdrawn after receiving escape therapy or completed treatment during 24weeks in CWP-TCZ301 study
* Patients who able to enroll in this study within 12 weeks after last infusion of CWP-TCZ301
* Willing to give written informed consent

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to Investigational product in CWP-TCZ301 study
* ALT or AST > ULNⅹ2.5
* Platelet count < 100ⅹ103/ μL
* WBC < 3,000/mm3
* Absolute neutrophil count < 1,000/mm3
* Absolute lymphocyte count < 500/mm3
* Total bilirubin > ULNⅹ2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety results | 48weeks
  1. All AE/ADR during study
  2. Physical examination including vital signs and ECG
  3. Clinical laboratory results

SECONDARY OUTCOMES:
Proportion of patients with ACR20, ACR50 and ACR70 responses at post therapy | 48weeks
Proportion of patients maintain with ACR20, ACR50 and ACR 70 responses at post therapy | 48weeks
Change of individual parameter in ACR core set | 48weeks
Change of individual parameter in DAS28 | 48weeks
Change of individual parameter in Rheumatoid factor | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univ. Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Choi IA, Sagawa A, Lee EY, Lee EB, Song YW. Tocilizumab Increases Body Weight and Serum Adipokine Levels in Patients with Rheumatoid Arthritis Independently of Their Treatment Response: a Retrospective Cohort Study. J Korean Med Sci. 2020 Jun 8;35(22):e155. doi: 10.3346/jkms.2020.35.e155. PMID 32508063